CLINICAL TRIAL: NCT02075632
Title: A Mult-Center, Open-Label Study to Evaluate Product Duration of Use Experience With Aclometasone Diproprionate Cream
Brief Title: Study to Evaluate Product Duration of Use Experience With Alclometasone Dipropionate Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2200440
Record Dates: First submitted 2014-01-28; First posted 2014-03-03 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Eczema; Allergy Symptoms; Psoriasis; Itch
Keywords: Alclometasone dipropionate; Eczema; Psoriasis; Itch
MeSH Terms: conditions — Eczema; Psoriasis; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alclometasone dipropionate cream (Experimental): Alclometasone dipropionate cream 0.05% will be applied by the participants topically on the affected areas per label instructions for 14 days.
  Interventions: Drug: Alclometasone dipropionate cream

INTERVENTIONS:
Drug: Alclometasone dipropionate cream — Alclometasone dipropionate cream 0.05% (15 g)

SUMMARY:
This is a multi-center, open-label study to evaluate whether participants follow the duration of use instructions for short-term use of alclometasone dipropionate in a population of participants with itchy skin conditions who would use OTC treatments for relief. The study population will be composed of two different cohorts: chronic condition sufferers (eczema or psoriasis) and participants who suffer from occasional itchy skin experiences (such as poison ivy, oak, sumac, insect bites, or skin irritations due to jewelry, cosmetics, detergents, or soaps) where an anti-itch medication would be used.

DETAILED DESCRIPTION:
Approximately 313 participants who are currently suffering from an itchy skin condition caused by eczema or psoriasis or any occasional itchy skin experiences will be enrolled into the study to get 250 participants who complete the study (at least 100 to each of the cohorts). After evaluation of the study criteria, the site staff will dispense product and a diary card to the subject to use over the next 14 days. At the end of the 14 days, each participant will come to the research site to return the remaining product and undergo the study termination interview with the Concentrics nurse via telephone. The study will be conducted in approximately 15 research sites located throughout the United States (US).

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 12 years of age.
* Condition: Currently experiencing itch associated with one of the following skin conditions:

  * psoriasis or eczema,
  * minor skin conditions such as those caused by poison ivy, oak, or sumac, insect bites, or use of cosmetics, soaps, detergents, or jewelry.
* Compliance: Subject or subject's parent or legal guardian understands and is willing, able and likely to comply with all study procedures and restrictions.
* Consent: Subject or subject's parent or legal guardian demonstrates ability to read and understand English and is willing to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form (and assent as appropriate).

Exclusion Criteria:

* Pregnancy: Women who are known to be pregnant (as self-reported) or who are intending to become pregnant over the duration of the study. Women of childbearing potential will be allowed to participate in the study so long as they are practicing a reliable method of contraception (e.g. hormonal birth control such as pill, patch, implant or injection; intrauterine device, double barrier methods, tubal ligation, vasectomized spouse or abstinence).
* Corticosteroid Use: Subject has used a corticosteroid treatment within two weeks of the screening visit at the start of the study.
* Breast-feeding: Women who are breastfeeding.
* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to alclometasone cream (or closely related compounds), or any of their stated ingredients.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit at the start of the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site
Pre-assignment Details: Participants with itchy skin conditions, who would use OTC treatments for relief
Groups:
- Chronic Condition: Participants who suffered from eczema or psoriasis where an anti-itch medication would be used.
- Occasional Itch: Participants who suffered from occasional itchy skin experiences (such as poison ivy, oak, sumac, insect bites, or skin irritations due to jewelry, cosmetics, detergents, or soaps) where an anti-itch medication would be used.
Period: Overall Study
Arm/Group | Chronic Condition | Occasional Itch
Started | 162 | 148
Completed | 161 | 143
Not Completed | 1 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Condition | Occasional Itch | Total
Number analyzed (Participants) | 162 | 148 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (15.68) | 50.6 (14.10) | 49 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 112 | 217
  Male | 57 | 36 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incorrect Duration of Use of the Medication
Description: Incorrect duration of use was defined as the use of study medication for more than 7 consecutive days and/or more than three times in a day. Participants were asked the reasons of doing so and they were allowed to select multiple reasons also, if applicable.
Time Frame: Day1-Day 14
Population: A participant was evaluable for analysis of the rate of incorrect use if he or she used the study medication at least once and provided use information at least 8 days after the enrollment visit.
Measure: Number; unit: Participants
Arm/Group | Chronic Condition | Occasional Itch
Number analyzed (Participants) | 161 | 143
Participants | 97 | 89

2. Secondary Outcome: Number of Times Per Day Participants Used the Product
Description: The number of study medication applications, was summarized for all subjects and by cohort in evaluable subjects.
Time Frame: Day1-Day14
Population: A subject was evaluable for average number of applications per day and maximum number of applications per day if he or she used the study medication at least once and provided use information at Visit 2. Data for four subjects was not available for this analysis.
Measure: Mean (Standard Deviation); unit: Applications
Arm/Group | Chronic Condition | Occasional Itch
Number analyzed (Participants) | 162 | 144
Applications
  Average Application Per Day | 1.95 (0.79) | 1.92 (0.65)
  Maximum Application Per Day | 2.6 (1.26) | 2.7 (1.05)

3. Secondary Outcome: Number of Days of Use
Description: The number of days subjects used the study medication was summarized for all subjects and by cohort in evaluable subjects.
Time Frame: Day 1-Day 14
Population: A subject was evaluable for summaries of number of days of use, if he or she used the study medication at least once and provided use information at Visit 2. Data for 4 subjects was not available for this analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Chronic Condition | Occasional Itch
Number analyzed (Participants) | 162 | 144
Days | 12.5 (2.70) | 11.8 (3.35)

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 48 hours after visit 2(14 days)
Description: The safety population included all subjects who used the study medication at least once and completed the Visit 2 study procedures, regardless of the time elapsed from enrollment to that visit. Out of 148 participants, 144 participants qualified for safety population in the occasional itch arm.
Arm/Group | Chronic Condition | Occasional Itch
Serious Adverse Events (participants affected / at risk) | 1/162 | 0/144
Other Adverse Events (participants affected / at risk) | 4/162 | 3/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Condition (N=162) | Occasional Itch (N=144)
Malignant Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Condition (N=162) | Occasional Itch (N=144)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.